CLINICAL TRIAL: NCT01399359
Title: A Study to Evaluate Different Decision-Making Approaches Used by Women Known to be at Increased Risk for Breast Cancer
Brief Title: Factors Influencing Decision-Making About the Use of Chemoprevention in Women at Increased Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NSABP-DMP-1; NSABP-DMP-1
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women who decide not to take a SERM: Women participate in the counseling session, questionnaire 1, and questionnaire 2, and the online questionnaire.
  Interventions: Behavioral: Counseling session; Other: Questionnaire 1; Other: Questionnaire 2; Other: online questionnaire
- Women who decide to take a SERM: Women participate in the counseling session, questionnaire 1 and questionnaire 2.
  Interventions: Behavioral: Counseling session; Other: Questionnaire 1; Other: Questionnaire 2

INTERVENTIONS:
Behavioral: Counseling session
Other: Questionnaire 1 — Questionnaire 1 assesses the recall and understanding of risk information given during the counseling session.
Other: Questionnaire 2 — Questionnaire 2 focuses on what factors, other thana the numerical risk-benefit analysis of SERM intake, are important in the decision-making process of women at increased risk for breast cancer.
Other: online questionnaire
  Groups: Women who decide not to take a SERM

SUMMARY:
RATIONALE: Learning about how patients make decisions about using chemoprevention may help doctors plan treatment in which more patients are willing to choose chemoprevention to reduce their breast cancer risk.

PURPOSE: This clinical trial studies factors influencing decision-making about the use of chemoprevention in women at increased risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To describe the influence of social, environmental, and psychological factors (sociality of medication intake, life-events, understanding of prevention, clinical situation) on the decision of women at risk for breast cancer as to whether or not to take chemoprevention agents.

Secondary

* To determine the implications of and influences on decision-making that a diagnosis of "being at risk for breast cancer" has for women.
* To determine what factors hinder women from taking chemoprevention for breast cancer.
* To field test a questionnaire that identifies the factors that influence the decision-making process of women at increased risk of breast cancer for whom chemoprevention is a medically indicated option.
* To describe the influence of social, environmental, and psychological factors on the decision of women at risk for breast cancer as to whether or not to take chemoprevention agents by menopausal status.
* For postmenopausal women who decide to take a selective estrogen-receptor modulator (SERM) for breast cancer prevention, to assess reasons for the choice of raloxifene versus tamoxifen.

OUTLINE: This is a multicenter study.

Participants undergo a counseling session about their increased risk for breast cancer and the use of a selective estrogen-receptor modulator (SERM), tamoxifen citrate or raloxifene, to reduce breast cancer risk. Some participants may have their counseling session video-recorded. They are also asked to review the video with their interviewers and to be contacted for a brief follow-up telephone interview.

Participants then complete an initial questionnaire to assess recall and understanding of risk information given to them during the counseling session. This first questionnaire is completed preferably on the same day of counseling before leaving the clinic or office. Participants also have the option to take the questionnaire home and return it to the study site within 2 weeks. Participants who return the first questionnaire complete a second one before leaving the clinic or office, or receive it by mail with a returned self-addressed stamped envelope. Participants who indicate on the second questionnaire that they do not want to take a SERM are asked to complete an online questionnaire. Participants who have not made a decision about SERM use within 3 months after counseling are contacted by telephone. They also receive the second questionnaire by mail 3 months after the telephone contact.

Interviewers, doctors, or other health-care professionals also complete questionnaires that indicate what was discussed during counseling sessions.

ELIGIBILITY:
Inclusion criteria

* The participant must be female.
* The participant must be greater than or equal to 35 years of age.
* The participant must be English-speaking.
* The participant must have been identified as being at increased risk for breast cancer as determined by the doctor/healthcare professional (HCP) . (Increased risk for breast cancer does not have to be based on a Gail score.)
* During the participant's counseling session, breast cancer risk and the use of SERMs for breast cancer risk reduction must have been discussed, as reported by the doctor/HCP who conducted the session. Note: This criterion does not apply to participants who are asked before the counseling session to participate in the video recording component of DMP-1 at the selected NSABP sites.

Exclusion criteria

* Previous invasive breast cancer of any type.
* Previous history of ductal carcinoma in situ (DCIS).
* Previous history of lobular carcinoma in situ (LCIS) if treated with mastectomy, radiation therapy, or endocrine therapy.
* Participation in any other cancer prevention study involving pharmacologic intervention(s) or osteoporosis prevention study involving pharmacologic intervention(s).
* Any history of or current tamoxifen, raloxifene, or other SERM therapy for any reason. (Participants are eligible if SERM use has been discussed prior to the counseling session as long as SERMs were never used.)

Ages: 35 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women at increased risk for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Social, environmental, and psychological influences on the decision of women at risk for breast cancer as to whether or not to take a SERM | Measured at start of study and at 3 to 6 months

SECONDARY OUTCOMES:
Factors hindering women from taking chemoprevention for breast cancer | Measured at start of study and at 3 to 6 months
Reasons for the choice of raloxifene vs tamoxifen among menopausal women | Measured at start of study and at 3 to 6 months
The implications of and influences on decision-making that a diagnosis of "being at risk for breast cancer" has for women. | Measured at start of study and at 3 to 6 months
To test a questionnaire that identifies the factors that influence the decision-making process of women at increased risk of breast cancer for whom chemoprevention is a medically-indicated option. | Measured at start of study and at 3 to 6 months
To describe the influence of social, environmental, and psychological factors on the decision of women at risk for breast cancer as to whether or not to take chemoprevention agents by menopausal status. | Measured at start of study and at 3 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Blakeslee SB, Gunn CM, Parker PA, Fagerlin A, Battaglia T, Bevers TB, Bandos H, McCaskill-Stevens W, Kennedy JW, Holmberg C. Talking numbers: how women and providers use risk scores during and after risk counseling - a qualitative investigation from the NRG Oncology/NSABP DMP-1 study. BMJ Open. 2023 Nov 19;13(11):e073138. doi: 10.1136/bmjopen-2023-073138. PMID 37984961
- [Derived] Gunn CM, Bokhour BG, Parker VA, Battaglia TA, Parker PA, Fagerlin A, McCaskill-Stevens W, Bandos H, Blakeslee SB, Holmberg C. Understanding Decision Making about Breast Cancer Prevention in Action: The Intersection of Perceived Risk, Perceived Control, and Social Context: NRG Oncology/NSABP DMP-1. Med Decis Making. 2019 Apr;39(3):217-227. doi: 10.1177/0272989X19827258. Epub 2019 Feb 25. PMID 30803311